CLINICAL TRIAL: NCT03376997
Title: An Open-Label, Randomized, Crossover Study to Evaluate Bioavailability of a Single 12 mg Dose of Perampanel for Three Intravenous Infusion Durations Relative to a Single 12 mg Perampanel Oral Tablet in Healthy Subjects
Brief Title: Study to Evaluate Bioavailability of a Single 12 mg Dose of Perampanel for Three Intravenous Infusion Durations Relative to a Single 12 mg Perampanel Oral Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: E2007-A001-050
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2017-12

CONDITIONS: Healthy Participants
Keywords: Bioavailability; Perampanel
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Perampanel: 30-minute IV infusion and 12 mg oral tablet (Experimental): Participants will be randomized on Day 1 of Treatment Period 1 to receive either a single 12 milligram (mg) dose of perampanel intravenous (IV) infusion (30-minute duration) or a single 12 mg oral tablet after an overnight fast. Participants will then receive the alternative treatment on Day 43 of Treatment Period 2. Drug administration will be separated by a washout of at least 6 weeks between the 2 treatment periods.
  Interventions: Drug: Perampanel
- Perampanel: 60-minute IV infusion and 12 mg oral tablet (Experimental): Participants will be randomized on Day 1 of Treatment Period 1 to receive either a single 12 mg dose of perampanel IV infusion (60-minute duration) or a single 12 mg oral tablet after an overnight fast. Participants will then receive the alternative treatment on Day 43 of Treatment Period 2. Drug administration will be separated by a washout of at least 6 weeks between the 2 treatment periods.
  Interventions: Drug: Perampanel
- Perampanel: 90-minute IV infusion and 12 mg oral tablet (Experimental): Participants will be randomized on Day 1 of Treatment Period 1 to receive either a single 12 mg dose of perampanel IV infusion (90-minute duration) or a single 12 mg oral tablet after an overnight fast. Participants will then receive the alternative treatment on Day 43 of Treatment Period 2. Drug administration will be separated by a washout of at least 6 weeks between the 2 treatment periods.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — IV infusion
  Other Names: E2007
Drug: Perampanel — Oral tablet
  Other Names: E2007

SUMMARY:
This study will be conducted to evaluate the bioavailability of a single 12 milligram (mg) dose of perampanel intravenous infusions of different durations relative to a single 12 mg dose of perampanel oral tablet in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, male or female, between 20 and 55 years of age (inclusive) at the time of informed consent
* Body mass index (BMI) of 18 to 32 kilograms per meters squared (kg/m^2) (inclusive) at Screening
* For Japanese participants:

  i. Born in Japan to Japanese parents and grandparents of Japanese descent; ii. Have been living outside Japan for less than 5 years; and iii. Lifestyle, including diet, has not changed significantly since leaving Japan
* Provide written informed consent
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Females of childbearing potential who:

  i. Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:
  1. total abstinence (if it is their preferred and usual lifestyle);
  2. an intrauterine device or intrauterine hormone-releasing system (IUS);
  3. a contraceptive implant;
  4. an oral contraceptive (with additional barrier method). Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation; or
  5. have a vasectomized partner with confirmed azoospermia ii. Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* Evidence of disease that may influence the outcome of the study within 4 weeks of dosing, eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or participants who have a congenital abnormality in metabolism
* Any history of gastrointestinal surgery that may affect pharmacokinetics (PK) profiles of perampanel, eg, hepatectomy, nephrectomy, digestive organ resection or any gastrointestinal procedure for the purpose of weight loss (including Lapband™), which would slow gastric emptying
* Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening or Baseline. A single repeat test for an abnormal vital sign and/or laboratory value is permitted, at the discretion of the Investigator.
* A prolonged QT/QTc interval (QTc >450 milliseconds [msec]) as demonstrated upon repeat ECG at Screening or Baseline
* Heart rate <50 or >100 beats per minute at Screening or Baseline
* History of ischemic heart disease (eg, acute coronary syndromes, stable angina), syncope or cardiac arrhythmias
* Systolic blood pressure >140 millimeters of mercury (mmHg) or <90 mmHg or diastolic blood pressure >90 mmHg or <60 mmHg at Screening or Baseline
* Hemoglobin <12.5 grams per deciliter (g/dL) or hematocrit ≤38% for males and postmenopausal females and hemoglobin <10 g/dL or hematocrit ≤33% for pre-menopausal females at Screening
* Participants who experienced a weight loss or gain of >10% between Screening and the first clinic check-in (Day -1)
* Participants who received blood products within 4 weeks, donated blood within 8 weeks, or donated plasma within 1 week of dosing
* Hypersensitivity to the study drug or any of its excipients
* Known severe or clinically significant history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
* Known to be human immunodeficiency virus (HIV) positive at Screening
* Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse within approximately the last 2 years or who have a positive urine drug, cotinine, or alcohol test at Screening or Baseline
* Engagement in strenuous exercise within 2 weeks before dosing (eg, marathon runners, weight lifters)
* Currently enrolled in another clinical trial or used any investigational drug or device within 30 days preceding informed consent
* Restrictions on prior and concomitant medications, food and beverages:

  i. Prescription drugs are prohibited within 4 weeks of dosing and over-the-counter (OTC) drugs within 2 weeks before dosing or throughout the Treatment Phase ii. Smoking or use of tobacco or nicotine-containing products is prohibited within 4 weeks before dosing and throughout the Treatment Phase iii. Intake of caffeinated beverages or food is prohibited within 72 hours before dosing and until 72 hours postdose iv. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect Cytochrome P450 (CYP) 3A4 enzyme or transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard] and charbroiled meats) is prohibited within 2 weeks before dosing and throughout the Treatment Phase v. Intake of herbal preparations containing St. John's Wort is prohibited within 4 weeks before dosing and throughout the Treatment Phase

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed concentration (Cmax) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (Day [D]1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  Cmax is the maximum plasma concentration of a drug after administration. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean value for area under the concentration versus time curve from time 0 to time of last measurable concentration (AUC[0-t]) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  AUC is a measure of actual body exposure to drug after administration of the drug. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean value for AUC versus time curve from time 0 to infinity (AUC[0-inf]) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  AUC is a measure of actual body exposure to drug after administration of the drug. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.

SECONDARY OUTCOMES:
Mean value for AUC versus time curve from time 0 to 72 hours (AUC[0-72h]) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  AUC is a measure of actual body exposure to drug after administration of the drug. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean time to reach maximum concentration (tmax) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  tmax is the time to reach maximum concentration following drug administration. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean terminal phase half-life (t1/2) postdose of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  t1/2 is the time required for the concentration of the drug to reach half of its original value. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean total clearance (CL) post intravenous (IV) infusion of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  CL is the volume of plasma cleared of drug per unit time. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Mean volume of distribution (Vd) post IV infusion of perampanel | predose; 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 (D1 and D43); 24 and 36 (D2 and D44); 48 (D3 and D45); 72 (D4 and D46); 120 (D6 and D48); 168 (D8 and D50); 336 (D15 and D57); and 504 (D22 and D64) hours after dosing start
  Vd is the apparent volume in which a drug is distributed. Dosing will occur on Day 1 of Treatment Period 1 and Day 43 of Treatment Period 2.
Number of participants with any treatment-emergent (TE) serious adverse event (SAE) | Up to approximately 16 weeks
  An SAE is any untoward medical occurrence that at any dose: results in death; is life threatening (an adverse event [AE] is considered life-threatening if, in the view of either the Investigator or Sponsor, its occurrence places the participant at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death.); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants with any non-serious TEAE | Up to approximately 16 weeks
  An AE is any untoward medical occurrence and does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product (IP), whether or not related to the IP. AEs include pre-existing conditions that worsen. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants with an abnormal, clinically significant laboratory parameter value | Up to approximately 16 weeks
  Clinical significance will be determined by the Investigator.
Number of participants requiring concomitant medication | Up to approximately 16 weeks
  Concomitant medications are medications that started after the date of the first dose of perampanel until the end of the study.
Number of participants with an abnormal, clinically significant vital sign value | Up to approximately 16 weeks
  Clinical significance will be determined by the Investigator.
Number of participants with an abnormal, clinically significant physical examination finding | Up to approximately 16 weeks
  Clinical significance will be determined by the Investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

REFERENCES:
- [Derived] Hussein Z, Majid O, Boyd P, Aluri J, Ngo LY, Reyderman L. Intravenous Perampanel as an Interchangeable Alternative to Oral Perampanel: A Randomized, Crossover, Phase I Pharmacokinetic and Safety Study. Clin Pharmacol Drug Dev. 2022 Jul;11(7):878-888. doi: 10.1002/cpdd.1107. Epub 2022 May 20. PMID 35596529